CLINICAL TRIAL: NCT06011889
Title: A Multicenter, Randomized, Double-blind Clinical Trial Evaluating the Efficacy and Safety of Etanercept Versus Placebo in the Treatment of Patients With SAPHO Syndrome
Brief Title: Study of the Efficacy and Safety of Etanercept Treatment in Patients With SAPHO Syndrome
Acronym: SAPHO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIGRIR_003SAPHO
Record Dates: First submitted 2023-07-28; First posted 2023-08-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: SAPHO Syndrome
MeSH Terms: conditions — Acquired Hyperostosis Syndrome | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etanercept (Experimental): treatment with etanercept in addition to NSAID treatment and/or classic Disease Modifying Antirheumatic Drugs
  Interventions: Drug: Etanercept
- Placebo (Placebo Comparator): treatment with placeboin addition to NSAID treatment and/or classic Disease Modifying Antirheumatic Drugs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — treatment with etanercept in addition to NSAID treatment and/or classic Disease Modifying Antirheumatic Drugs
  Arms: Etanercept
Drug: Placebo — treatment with placebo in addition to NSAID treatment and/or classic Disease Modifying Antirheumatic Drugs
  Arms: Placebo

SUMMARY:
The study includes adult patients with SAPHO syndrome (ORPHA: 793), meeting the modified classification criteria according to Kahn (2003), with the ineffectiveness of standard treatment (patient's global assessment of the disease on the VAS scale greater than or equal to 4 cm with accompanying pain on the VAS scale greater than or equal to 4 cm) treated with non-steroidal anti-inflammatory drugs in a stable dose for at least 4 weeks and/or classical disease-modifying antirheumatic drugs in stable doses for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SAPHO syndrome according to modified Kahn criteria from 2003.
2. Age over 18.
3. Patient overall disease and pain assessment on VAS both ≥ 4 cm.
4. Expressing informed consent to participate in the study.

Exclusion Criteria:

1. According to the Summary of Product Characteristics (SmPC) for Enbrel.
2. Pregnancy, breastfeeding, inability to use effective contraception during the examination.
3. Change in the dose of NSAIDs treatment in the last 4 weeks.
4. Dose modification of disease-modifying antirheumatic drugs (DMARDs) over the past 12 weeks.
5. Use of biological drugs / synthetic targeted drugs in the last 12 weeks.
6. Use of corticosteroids (orally or local injections), bisphosphonates and/or antibiotics in the last 4 weeks.
7. Any medical condition that the investigator judges to contraindicate etanercept treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-10-18 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in the scope of disease activity as assessed by the patient- a decrease in the overall disease activity on the Visual Analogue Scale by min. 50 percent and a decrease in pain assessed by the patient on the Visual Analogue Scale by min. 50 percent | 12 weeks (day 85)
  Change in the scope of disease activity as assessed by the patient - a decrease in the overall disease activity as assessed by the patient on the Visual Analogue Scale by min. 50 percent after 12 weeks from randomization day and a decrease in pain assessed by the patient on the Visual Analogue Scale by min. 50 percent after 12 weeks from randomization day. The minimum value is - 0, and the maximum value is - 100 mm. The higher scores mean a worse outcome. A decrease by a minimum of 50 percent means a better outcome.

SECONDARY OUTCOMES:
Change in patient-assessed disease activity | after 4 and 8 weeks
  Change in patient-assessed disease activity - a minimum 50 percent decrease in patient-assessed Visual Analogue Scale overall disease activity from the randomization score at weeks 4 and 8 and a minimum 50 percent decrease in patient-assessed Visual Analogue Scale pain from the score on daily basis randomization after 4 and 8 weeks. The minimum value is - 0, and the maximum is - 100 mm. The higher scores mean a worse outcome. A decrease by a minimum of 50 percent means a better outcome.
Occurrence of remission | after 4, 8 and 12 weeks
  Occurrence of remission - complete resolution of osteoarticular and skin complaints in the patient's assessment - after 4, 8 and 12 weeks from randomization day
Occurrence of partial remission | after 4, 8 and 12 weeks
  Occurrence of partial remission - complete resolution of osteoarticular or skin symptoms in the patient's assessment - after 4, 8 and 12 weeks from randomization day
Occurrence of the patient acceptable symptom state (PASS score) | after 4, 8 and 12 weeks
  Occurrence of the patient acceptable symptom state (PASS score) after 4, 8 and 12 weeks from randomization day. Possible answer- "yes" or "no", with "yes" means a better outcome.
Change in physician-assessed disease activity | at 4, 8 and 12 week
  Improvement in physician-assessed disease activity - a minimum 50 percent decrease in physician-assessed overall disease activity on the Visual Analogue Scale from the randomization score at 4, 8 and 12 weeks. The minimum value is - 0, and the maximum is - 100 mm. The higher scores mean a worse outcome. A decrease by a minimum of 50 percent means a better outcome.
Change in the C-reactive Protein from Randomization Day Score | at Weeks 4, 8 and 12
  Change in C-reactive Protein from Randomization Day Score at Weeks 4, 8 and 12. A decrease in C-reactive Protein means improvement.
Change in the Erythrocyte Sedimentation Rate from Randomization Day Score | at Weeks 4, 8 and 12
  Change in the Erythrocyte Sedimentation Rate Score from Randomization Day Score at Weeks 4, 8 and 12. A decrease in the Erythrocyte Sedimentation Rate Score means improvement.
Change in quality of life on the Short Form-36 health survey | at 4, 8 and 12 weeks
  Change in quality of life on the Short Form -36 (SF-36) health survey from the score on the day of randomization at 4, 8 and 12 weeks. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Change in the Work Productivity and Activity Impairments (WPAI) from the Randomization Day Score | after 4, 8 and 12 weeks
  Change in the Work Productivity and Activity Impairments (WPAI) from the Randomization Day Score after 4, 8 and 12 weeks. WPAI contains four domains. For each domain, the minimum value is 0 percent, and the maximum is 100 percent. Decreased Work Productivity and Activity Impairments (WPAI) Score means improvement.
decrease in Ankylosing Spondylitis Disease Activity Score (ASDAS- C-reactive protein) ≥1.1 | after 4, 8 and 12 weeks
  In patients with axial involvement, a decrease in Ankylosing Spondylitis Disease Activity Score (ASDAS- C-reactive protein) ≥1.1 from the Randomization Day Score at weeks 4, 8, and 12. The minimum value is 0, the maximum value is infinity. A decrease means a better outcome.
a decrease in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score of at least 50 percent | after 4, 8 and 12 weeks
  a decrease in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score of at least 50 percent from the Randomization Day Score at weeks 4, 8, and 12 was achieved (applies to patients with axial involvement). The minimum value is 0, the maximum value is 10. A decrease by a minimum of 50 percent means a better outcome.
status of remission- Ankylosing Spondylitis Disease Activity Score (ASDAS- C-reactive protein) below 1.3 | after 4, 8 and 12 weeks
  status of remission - Ankylosing Spondylitis Disease Activity Score (ASDAS- C-reactive protein) below 1.3 - after 4, 8 and 12 weeks from randomization day (applies to patients with axial involvement). A score below 1.3 means a better outcome.
decrease in the Bath Ankylosing Spondylitis Functional Index (BASFI) by a minimum of 50 percent | after 4, 8 and 12 weeks
  a decrease in the Bath Ankylosing Spondylitis Functional Index (BASFI) by a minimum of 50 percent compared to the result on the day of randomization after 4, 8 and 12 weeks (applies to patients with axial involvement). The minimum value is 0, the maximum value is 10. A decrease by a minimum of 50 percent means a better outcome.
decrease in the Dermatology Life Quality Index (DLQI) by at least 50 percent from the result on the day of randomization | after 4, 8 and 12 weeks
  In patients with severe acne - a decrease in the Dermatology Life Quality Index (DLQI) by at least 50 percent from the result on the day of randomization after 4, 8 and 12 weeks. The minimum value is 0, the maximum value is 30. The decrease by a minimum of 50 percent means a better outcome.
decrease in Body Surface Area (BSA) index by a minimum of 50 percent from the score on the day of randomization after 4, 8 and 12 weeks | after 4, 8 and 12 weeks
  For patients with psoriasis: decrease in Body Surface Area (BSA) index by a minimum of 50 percent from the score on the day of randomization after 4, 8 and 12 weeks. The minimum value is 0 percent, and the maximum value is 100 percent. The decrease by a minimum of 50 percent means a better outcome.
decrease in the Dermatology Life Quality Index (DLQI) by a minimum of 50 percent | after 4, 8 and 12 weeks
  For patients with psoriasis: decrease in the Dermatology Life Quality Index (DLQI) by a minimum of 50 percent from the score on the day of randomization after 4, 8 and 12 weeks. The minimum value is 0, the maximum value is 30. The decrease by a minimum of 50 percent means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Wroński, PhD, MD, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation
Locations (1):
- Centrum Wsparcia Badań Klinicznych, Warsaw, Masovian Voivodeship, Poland